CLINICAL TRIAL: NCT01528566
Title: Effect of Tai Chi on Osteoarthritic Knee Pain in Elders With Mild Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21NR01003
Record Dates: First submitted 2012-01-24; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Osteoarthritis, Knee; Dementia
Keywords: osteoarthritis, knee; Cognitive impairment; Tai Chi
MeSH Terms: conditions — Osteoarthritis, Knee; Dementia; Cognitive Dysfunction | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi (Experimental)
  Interventions: Behavioral: Tai Chi
- Attentation control (Placebo Comparator)
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: Tai Chi — The experimental group received three sessions of Sun Tai Chi (TC) a week for 20 weeks (20-to-40 minute exercise plus a 5-minute rest per session). Sun TC includes 6 basic and 6 advanced forms designed for all ages with arthritis seeking a joint-safe exercise routine.
  Arms: Tai Chi
Behavioral: Attention control — The attention control group participated in health education, culture related activities and other activities for a total of 20 weeks. The attention control protocol was standardized in terms of teaching content, materials and duration. The length and frequency of the activities carried out in this group closely matched those in the TC group.
  Arms: Attentation control

SUMMARY:
This is the first study to test the effect of Tai Chi on pain from knee osteoarthritis in community-dwelling elders with mild cognitive impairment. If Tai Chi is effective in reducing pain, clinicians can use it routinely with this population; then elders can maintain their functional ability longer, and perhaps delay or prevent long-term care admission, and the investigators can save health care dollars.

DETAILED DESCRIPTION:
Up to 33% of all elders and 40% of elders over age 70 experience knee osteoarthritis (OA), a leading cause of pain and disability. Further, up to 15.3% of elders age 65 have CI, and the prevalence of cognitive impairment (CI) doubles every 5 years after age 65. The prevalence of OA in elders with CI is comparable to that in elders without CI. Cognitive impairment limits elders' ability to perform daily activities, and their functional capacity declines more rapidly than in elders without CI. Having knee OA pain in addition to CI further limits elders' activities. Without proper treatment of knee OA pain, elders with CI may avoid basic daily activities, such as rising, walking, standing, and climbing stairs because these aggravate pain. By avoiding these basic activities, they gradually lose muscle strength, range of motion, and mobility, which leads to further physical deconditioning and social isolation. With aging of the baby boomers and advances in health care, the number of elders with both CI and OA will increase fourfold by 2050. Alleviating knee pain in elders with CI and knee OA could preserve their functioning, perhaps delay institutionalization, and save healthcare dollars. Since pharmacological interventions produce serious side effects and inadequately reduce pain, especially in elders with CI, adjuncts such as Tai Chi (TC) are needed. A low-impact aerobic exercise, TC involves slowly stretching the limbs and trunk and ultimately re-establishes normal mechanics of the knee joints, which reduces knee OA pain. The United States Arthritis Foundation and the American Geriatrics Society have endorsed TC to reduce knee OA pain; but no study has investigated the effect of TC on knee OA pain in elders with CI. The primary aims of this study are:

1. To test the efficacy of a modified TC program in reducing knee OA pain in community-dwelling elders with mild CI.
2. To test the efficacy of a modified TC program in improving physical function and quadriceps strength.
3. To investigate feasibility and compliance issues in conducting TC.
4. To estimate the clinical significance of TC for pain reduction in community dwelling elders with mild CI.

The results of this study will help us design a full-scale RCT with a precise estimate of the sample size and dosage of TC needed for reducing knee OA pain in community-dwelling elders with mild CI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years or order;
2. A MMSE score of 18-28;
3. Diagnosis of knee OA based on medical history reviewed with elders or family members/staff and confirmation from the physician/APN;
4. Self-report of knee OA pain ≥ 2 on the VDS, or pain score ≥ 3 on the WOMAC pain subscale;
5. Ability to speak English;
6. Physician's/APN's permission to participate;
7. No regular exercise program in the past month;
8. Ambulation without assistance from staff or a walking device for 50 meters; and
9. Ability to stand and maintain balance for 1 minute without a walking device

Exclusion Criteria:

1. Uncorrectable moderate or severe hearing or vision deficits;
2. Parkinson's disease;
3. Cancer pain;
4. Chronic pain conditions, such as rheumatoid arthritis, fibromyalgia, or severe low back pain;
5. Diabetic neuropathy;
6. Arthroscopic surgery or total knee- or hip-replacement surgery in the past 6 months;
7. Fractures in the past 6 months;
8. Major psychiatric disorder or positive screen for depressive symptoms (GDS-15 score ≥ 5) without taking medication;
9. History of falls in the past 3 months; or
10. Vertigo in the past month

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain at Week 5 | Week 5
  Measured by 1). the WOMAC pain subscale; 2). the Verbal Descriptor Scale (VDS); 3). Keefe observational method; and 4). Analgesic intake.
Change from baseline in pain at Week 9 | Week 9
  Measured by 1). the WOMAC pain subscale; 2). the Verbal Descriptor Scale (VDS); 3). Keefe observational method; and 4). Analgesic intake.
Change from baseline in pain at Week 13 | Week 13
  Measured by 1). the WOMAC pain subscale; 2). the Verbal Descriptor Scale (VDS); 3). Keefe observational method; and 4). Analgesic intake.
Change from baseline in pain at Week 17 | Week 17
  Measured by 1). the WOMAC pain subscale; 2). the Verbal Descriptor Scale (VDS); 3). Keefe observational method; and 4). Analgesic intake.
Change from baseline in pain at Week 21 | Week 21
  Measured by 1). the WOMAC pain subscale; 2). the Verbal Descriptor Scale (VDS); 3). Keefe observational method; and 4). Analgesic intake.

SECONDARY OUTCOMES:
Physical function | Week 1 (baseline), week 5, week 9, week 13, week 17 and week 21 (post-test) for a total of 6 time points
  Measured by 1). WOMAC Physical Function subscale; and 2). Get Up and Go (GUG)
Cognitive function | Week 1 (baseline), week 5, week 9, week 13, week 17 and week 21 (post-test) for a total of 6 time points
  Mini Mental Status Exam (MMSE)
Stiffness | Week 1 (baseline), week 5, week 9, week 13, week 17 and week 21 (post-test) for a total of 6 time points
  WOMAC Stiffness subscale
Quadriceps strength | Week 1 (baseline), week 5, week 9, week 13, week 17 and week 21 (post-test) for a total of 6 time points
  Measured by the Sit-To-Stand (STS)
Pain level (each session) | Participants will be followed for the duration of intervention period (20 weeks)
  Measured by the Verbal Descriptor Scale (VDS)

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Feng Tsai, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical asciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Tsai PF, Chang JY, Chowdhury N, Beck C, Roberson PK, Rosengren K. Enrolling older adults with cognitive impairment in research: lessons from a study of Tai Chi for osteoarthritis knee pain. Res Gerontol Nurs. 2009 Oct;2(4):228-34. doi: 10.3928/19404921-20090731-03. Epub 2009 Oct 27. PMID 20077977
- [Derived] Tsai PF, Chang JY, Beck C, Kuo YF, Keefe FJ, Rosengren K. A supplemental report to a randomized cluster trial of a 20-week Sun-style Tai Chi for osteoarthritic knee pain in elders with cognitive impairment. Complement Ther Med. 2015 Aug;23(4):570-6. doi: 10.1016/j.ctim.2015.06.001. Epub 2015 Jun 9. PMID 26275650
- [Derived] Tsai PF, Chang JY, Beck C, Kuo YF, Keefe FJ. A pilot cluster-randomized trial of a 20-week Tai Chi program in elders with cognitive impairment and osteoarthritic knee: effects on pain and other health outcomes. J Pain Symptom Manage. 2013 Apr;45(4):660-9. doi: 10.1016/j.jpainsymman.2012.04.009. Epub 2012 Sep 24. PMID 23017610